CLINICAL TRIAL: NCT02395874
Title: MP-LoGa: Bi-hemispheral Transcranial Direct Current Stimulation to Improve the Severe Aphasia in Subacute Stroke Patients: a Randomized, Placebo-controlled, Double Blinded Multi-center Trial
Brief Title: tDCS and Speech Therapy to Improve Aphasia
Acronym: MP-LOGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Park AG (Industry)
Responsible Party: Principal Investigator, Cordula Werner, Head of Research Lab, Medical Park AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-LOGA
Record Dates: First submitted 2015-03-11; First posted 2015-03-24 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Aphasia, Global; Stroke; Transcranial Direct Current Stimulation; Speech Therapy
MeSH Terms: conditions — Aphasia; Stroke; Communication Disorders | interventions — Transcranial Direct Current Stimulation; Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- verum-tDCS (Experimental): verum-tDCS+ speech therapy
  Interventions: Procedure: tDCS + speech therapy
- sham-tDCS (Sham Comparator): sham-tDCS + speech therapy
  Interventions: Procedure: tDCS + speech therapy

INTERVENTIONS:
Procedure: tDCS + speech therapy — Patients either receive 20min of tDCS with 2mA + speech therapy every work for 6 weeks. The anodal electrode will be placed either on the homologous speech area (TACS) in the right hemisphere or on the speech area perilesional in the left hemisphere (PACS). The cathodal electrode will be placed contralateral. Patients in group B will follow the same protocol, except for the stimulation intensity (2 mA versus 0 mA) the speech therapist will apply the tdcs according to the protocol. The tdcs machine is out of sight of the patient, so that she/he does not see, whether the machine is switched on or not. In case of sham stimulation the device will be switched on very slowly for the first 20 s and will than be set back to 0mA within the following 10 s. So that the patient will feel also the characteristic tingling under the electrodes.

SUMMARY:
To study the effect of combined tDCS plus speech therapy compared to sham-tDCS plus speech therapy in subacute stroke patients suffering from moderate or severe aphasia. The patients will be randomized by a computer-generated lot. Assessment will be performed at study onset, after six weeks at the end of the specific intervention and 4 months after stroke onset for follow-up.

DETAILED DESCRIPTION:
Approximately 25% of all patients after stroke suffer from aphasia. The aphasia could be so severe, that the patient cannot produce any words at all, and so the communication ability is rather poor. In that case speech therapy is the most common therapy, but the functional outcome for the patient is often not sufficiently. The transcranial direct current stimulation (tDCS) might improve the outcome of speech therapy in patients with severe aphasia. The patients will be randomized either to verum stimulation (group A) or sham stimulation (group B). In group A they will receive every workday for 6 weeks 20min of tDCS with 2 mA in combination with a 30 min speech therapy. In group B they will receive every workday for 6 weeks 20min of tDCS with 0 mA in combination with a 30 min speech therapy. The anodal electrode will be placed in case of a total anterior circulation stroke on the homologous speech area on the right hemisphere and in case of a partial anterior circulation stroke perilesional on the left hemisphere. The cathode will be positioned contralateral.

ELIGIBILITY:
Inclusion Criteria:

* first time stroke (ischemic or hemorrhagic), either with a total or partial anterior circulation stroke according to the Bamford classification
* stroke interval 10-45 days
* moderate or severe aphasia, i.e. Goodglass-Kaplan-Communication-Scale (GKS, 0,1 or 2)
* native speaker - german
* age 18-90

Exclusion Criteria:

* other neurological diseases affecting the CNS
* known history of epileptic fits, except for an immediate fit
* signs in the EEG of increased cortical excitability
* patients with hemicraniectomy
* fluent aphasia, i.e. GKS 3,4 or 5
* speech apraxia
* reduced sensibility of the scalp
* previously radiated scalp
* metallic parts or implants in the brain
* participation in other interventional studies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Goodglass-Kaplan communication scale (GKS, 0-5) | 10-15 min
  the GKS is an ordinal scale, which assesses the communication ability of the patient from 0 to 5.
Aphasia Check-list (ACL, 0-148) | 30-45 min
  a german tool to assess language (analogous to the Aachener Aphasie Test). it measures a) colour-figure test, b) word generation and c) single speech domains

SECONDARY OUTCOMES:
Aphasic depression rating scale (ADRS, 0-32) | 5 min
  rates the depression in patients with aphasia
Alterskonzentrationstest (AKT, 0-35) | 5 min
  assesses the concentration and vigilance of elderly people with stroke
Barthel-Index (BI,0-100) | 5min
  evaluates the activities of daily living in patients suffering from stroke
Rivermead Motor Assessment - Arm (RMA, 0-15) | 5-10 min
  assesses the motor control of the upper extremity in patients with stroke

OTHER OUTCOMES:
Electroencephalography (EEG) | 30min
  to record spontaneous brain activity and to exclude increased cortical excitability

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Hesse, Prof. Dr., Principal Investigator — Medical Park Berlin, Charité - University Medicine Berlin
Locations (1):
- Medical Park Berlin Humboldtmuehle, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Hesse S, Waldner A, Mehrholz J, Tomelleri C, Pohl M, Werner C. Combined transcranial direct current stimulation and robot-assisted arm training in subacute stroke patients: an exploratory, randomized multicenter trial. Neurorehabil Neural Repair. 2011 Nov-Dec;25(9):838-46. doi: 10.1177/1545968311413906. Epub 2011 Aug 8. PMID 21825004
- [Result] Polanowska KE, Lesniak M, Seniow JB, Czlonkowska A. No effects of anodal transcranial direct stimulation on language abilities in early rehabilitation of post-stroke aphasic patients. Neurol Neurochir Pol. 2013 Sep-Oct;47(5):414-22. doi: 10.5114/ninp.2013.38221. PMID 24166562